CLINICAL TRIAL: NCT00657865
Title: Gene Expression Profiling in Skeletal Muscle of Healthy Subjects Treated With Ramipril
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Markus Mueller, Prof. Dr, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Ram_Gep_1; 2007-007276-41
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
MeSH Terms: interventions — Ramipril

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Ramipril
  Interventions: Drug: ramipril
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ramipril — oral intake
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
This project investigates the effect of ACE-inhibition on cellular metabolism by gene expression profiling of human muscle tissue, obtained by biopsy prior to and after ramipril intake.

This should contribute to our understanding of the pathomechanisms involved in diabetes and the clinical effect of ACE-inhibition on patients with diabetes/metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Healthy defined as absence of relevant disease
* Caucasian
* Aged 18-45 years
* BMI: 18-28 kg/m2
* Signed informed consent
* Blood pressure between 110/45 and <140/90 (twice at screening)

Exclusion Criteria:

* History of renal artery stenosis

  * angioneurotic edema
  * psoriasis
  * relevant renal diseases
* RR at screening < 110/45 mmHg.
* Diabetes, history of hypertension, RR > 140/90 at screening, cardiovascular disease
* Known Diabetes mellitus of parents
* HIV or Hepatitis B/C positive virology
* Allergy or hypersensitivity against ACE-inhibitors / ramipril or to xylocain
* Contraindications against the use of the drug according to the SmPC, history of angioedema
* Any drug intake 3 weeks prior to first study day
* History of excessive bleeding tendency / hemophilia
* Presence of relevant illness within the last 3 weeks
* Suspected non-compliance with study instructions and life-style requirements
* Alcohol or drug abuse
* Blood/Plasma donation within 4 weeks prior to study day
* Previous exposure to antihypertensive drugs, ACE-inhibitors, in particular ramipril
* Current smoking (any quantity), (at least 6 months of non-smoking required)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Genome-wide gene expression measurements in skeletal muscle at baseline and in response to ramipril intake. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Markus Mueller, MD, Principal Investigator — Medical University of Vienna, Dep. of Clinical Pharmacology
Locations (1):
- Medical University Vienna, Department of Clinical Pharacology, Vienna, Vienna, Austria